CLINICAL TRIAL: NCT02001818
Title: Phase II Study of Nilotinib Plus Pegylated Interferon Alfa-2b as First-line Therapy in Chronic Phase Chronic Myelogenous Leukaemia Aiming to Maximize Complete Molecular Response and Major Molecular Response.
Brief Title: Pegylated Interferon Alfa-2b and Nilotinib for Augmentation of Complete Molecular Response in Chronic Myeloid Leukaemia
Acronym: PInNACLe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Leukaemia and Lymphoma Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML11; ACTRN12612000851864 (Other: ANZCTR)
Record Dates: First submitted 2013-11-12; First posted 2013-12-05 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Chronic Myeloid Leukaemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; peginterferon alfa-2b; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib or Imatinib with Peginterferon (Experimental): Nilotinib 300mg twice daily for 24 months. Pegylated interferon alpha-2b 30-50 micrograms subcutaneously once weekly for maxium 21 months (3 months after trial registration).
  Patients intolerant of nilotinib may be switched to appropriate doses of imatinib
  Interventions: Drug: Nilotinib, Pegylated interferon alpha-2b, Imatinib

INTERVENTIONS:
Drug: Nilotinib, Pegylated interferon alpha-2b, Imatinib — All patients joining the study will receive treatment with oral nilotinib at 300mg twice daily. This will be given as monotherapy for 3 months initially, prior to commencement of combination therapy with Pegylated interferon alpha-2b added to nilotinib. Patients intolerant of nilotinib will have the option of switching to imatinib.

SUMMARY:
The treatment of CML and the expected survival has been revolutionised since the introduction of tyrosine kinase inhibitors (TKIs) such as nilotinib. Despite their effectiveness, these drugs will never totally remove CML affected cells from the body. In order to achieve this goal, and potentially enable CML patients to live without the daily need for TKIs, other features of the patient's immune system may need to be harnessed. One possibility is using externally administered interferon (IFN) to augment the response induced by the TKI.

This study will assess the response in terms of length of survival, detection of minimal disease levels and time until disease worsens in patients with chronic phase CML who are taking nilotinib and pegylated Interferon. Patients will commence taking nilotinib for 3 months, and once tolerated, will simultaneously be treated with injected pegIFN for up to 2 years. Patients can continue taking nilotinib beyond this time providing they are receiving benefit. Options are available for patients to decrease or increase their dose or to switch to another TKI, imatinib, to ensure a balance between drug effectiveness and minimal side effects is achieved.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be satisfied for enrolment in the study.

1. Post-pubertal male or female patients aged 18 years or above.
2. Newly diagnosed (within Three months of study entry) Ph+ CML-Chronic Phase with a quantifiable "breakpoint cluster region - Abelson murine leukemia" (BCR-ABL) transcript
3. No prior therapy for CML and no other current anti-leukaemic therapies (other than prior or current treatment with hydroxyurea or anagrelide).
4. No signs of extramedullary leukaemia, except for hepatosplenomegaly.
5. Documented chronic-phase CML as defined by:

   i. <15% blasts in both the peripheral blood and bone marrow ii. <30% blasts and promyelocytes in both the peripheral blood and bone marrow iii. <20% basophils in the peripheral blood iv. Platelet count >100 × 109/L (Note: Patients will be considered to be in chronic phase if their platelet count is ≤ 100 x 109/L as a result of treatment with hydroxyurea or anagrelide provided that all of the other criteria for chronic phase CML are met).
6. Eastern Cooperative Oncology Group Performance Status score ≤2 (see Appendix 2)
7. Patients must have the following laboratory values:

   1. Potassium level > Lower Limit of Normal (LLN)
   2. Calcium (corrected for serum albumin) > Lower Limit of Normal (LLN)
   3. Magnesium level > Lower Limit of Normal (LLN)
   4. Phosphorus > Lower Limit of Normal (LLN)
   5. ALT and AST < 2.5 × ULN or < 5.0 × Upper limit of normal (ULN) if considered due to tumour
   6. ALP < 2.5 × Upper limit of normal (ULN) unless considered due to tumour
   7. Bilirubin < 1.5 × Upper limit of normal (ULN) unless due to Gilbert's syndrome
   8. Creatinine < 1.5 × Upper limit of normal (ULN)
   9. Amylase and lipase < 1.5 × Upper limit of normal (ULN) Note: Biochemical abnormalities that resolve after corrective measures pose no impediment to re-screening.

a) Female patients of childbearing potential must have a negative serum pregnancy test within one week prior to study entry OR have been amenorrhoeic for at least 12 months.

b) All patients of reproductive potential must agree to use birth control for the duration of the study. This is only required for as long as the patient has reproductive potential. The type of birth control is a decision which should be made between the treating clinician and the patient.

9.Life expectancy of more than 12 months. 10.Patient has given written, informed consent to participate in the study (which includes consent to obtain samples for the correlative study except in a rare case where a site does not have the capacity to participate in the correlative study).

Exclusion Criteria:

Presence of any of the following criteria will exclude the subject from enrolment in the study.

1. Patients who have previously received radiotherapy to >25% of their bone marrow.
2. Patients who have undergone major surgery within the 4 weeks prior to study entry or have not recovered from earlier surgery.
3. Impaired cardiac function, including any of the following:

   1. Inability to monitor the QT/corrected QT intervak (QTc) interval on ECG
   2. Long QT syndrome or a known family history of long QT syndrome.
   3. Resting bradycardia (<50 beats per minute) suspected to be secondary to cardiac pathology
   4. QTc > 450 msec on baseline ECG (using the QTc formula). If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
   5. Other clinically significant uncontrolled heart disease (e.g. congestive heart failure or uncontrolled hypertension)
   6. History of or presence of clinically significant ventricular or atrial tachyarrhythmias, including atrial fibrillation
4. History of arterial vascular disease including coronary artery disease (Angina, myocardial infarction), cerebrovascular disease (Transient ischaemic attacks and strokes), peripheral vascular disease, retinal artery thromboses and mesenteric arterial thromboses.
5. Treatment with agents (other than warfarin) that prolong QT interval or inhibit Cytochrome P450 3A4 (CYP3A4), unless judged to be clinically essential.
6. Another primary malignant disease, except for such conditions that do not currently require treatment, lesions that can be or had been completely excised (eg Skin Cancers) and neoplasms that does not significantly affect long term survival of the patient
7. Significantly impaired GI function or GI disease that may alter nilotinib absorption.
8. Other concurrent uncontrolled medical conditions (e.g. uncontrolled diabetes, uncontrolled or unstable thyroid disease, active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol.
9. History of confirmed acute or chronic pancreatitis.
10. Cytopathologically confirmed Central Nervous System(CNS) infiltration. [In the absence of suspicion of CNS involvement, lumbar puncture is not required.]
11. Patients unwilling or unable to comply with protocol and patients with a history of noncompliance or inability to grant informed consent.
12. Known diagnosis of human immunodeficiency virus (HIV) infection.
13. Prior allogeneic stem cell transplantation
14. Patients who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Male and female patients of childbearing potential must agree to employ an effective method of birth control throughout the study. The type of birth control is a decision which should be made between the treating clinician and the patient
15. Known history of uncontrolled depression or any other psychiatric disease likely to be exacerbated by study treatment. A formal psychiatric assessment at baseline is not required.
16. Current participation in another therapeutic clinical trial (participation in clinical trials that do not involve active interventions is not an exclusion for the study.)
17. Previous adverse reaction to the trial drug/s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
level of BCR-ABL | 24 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tim Hughes, MBBS, MD, FRACP, FRCPA, Principal Investigator — Royal Adelaide Hospital; Andrew Grigg, MBBS, MD, FRACP, FRCPA, Principal Investigator — Austin Hospital, Melbourne Australia; David Yeung, BSc(Med), MBBS(Hons),FRACP, Principal Investigator — SA Pathology
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia